CLINICAL TRIAL: NCT05536349
Title: Time-limited Triplet Combination of Pirtobrutinib, Venetoclax, and Obinutuzumab for Patients With Treatment-naïve Chronic Lymphocytic Leukemia (CLL) or Richter Transformation (RT)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Loxo Oncology, Inc. (Industry); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0578; NCI-2022-07625 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — pirtobrutinib; obinutuzumab; venetoclax; Valacyclovir; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pirtobrutinib plus Venetoclax plus Obinutuzumab (combination) (Experimental): Participants will receive the study drugs in cycles. Each cycle is 28 days.
  Interventions: Drug: Pirtobrutinib; Drug: Obinutuzumab; Drug: Venetoclax; Drug: Valacyclovir; Drug: Allopurinol

INTERVENTIONS:
Drug: Pirtobrutinib — Given by PO
Drug: Obinutuzumab — Given by (IV) vein
  Other Names: GA101; Gazyva; RO5072759
Drug: Venetoclax — Given by PO
  Other Names: ABT-199; GDC-0199
Drug: Valacyclovir — Given by PO
Drug: Allopurinol — Given by PO

SUMMARY:
To learn if the combination of pirtobrutinib (also called LOXO-305), venetoclax, and obinutuzumab is safe and effective when given to patients with chronic lymphocytic leukemia (CLL) or Richter transformation (RT) who have not previously received treatment.

DETAILED DESCRIPTION:
Primary Objective:

1. Estimate the therapeutic activity (undetectable measurable residual disease [U-MRD] rate) of combined pirtobrutinib, venetoclax, and obinutuzumab in patients with previously untreated CLL/SLL (cohort 1) by undetectable measurable residual disease (U-MRD) rate and Richter transformation (cohort 2) by overall response rate (ORR) (defined as CMR//PMR).

Secondary Objectives:

1. To estimate the therapeutic activity of combination therapy by determining:

   1. Combined response rate (defined as CR/CRi/PR) as assessed by the investigator for cohort 1 (CLL/SLL)
   2. Progression free survival (PFS) and overall survival (OS).
   3. U-MRD response with next generation sequencing assay for cohort 2
2. To determine the safety and tolerability of this combination therapy

Exploratory Objective:

1. To study immunological and molecular changes in the peripheral blood and bone marrow in response to pirtobrutinib, venetoclax, and obinutuzumab.
2. To evaluate the kinetics of MRD response over time

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of previously untreated CLL/SLL meeting iwCLL 2018 indication for treatment (cohort 1) or with a diagnosis of previously untreated or relapsed/refractory RT arising from CLL (cohort 2). Previously untreated patients with RT must have received prior therapy for CLL.
2. At least 18 years of age
3. Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2
4. Adequate hepatic function

   1. Total bilirubin ≤1.5 x upper limit of normal (ULN) or ≤3 x ULN for patients with Gilbert's disease or documented disease involvement of liver (In pts with elevated total bilirubin due to increased indirect bilirubin, pts with direct bilirubin ≤1.5 x ULN are eligible)
   2. ALT and AST ≤3.0 x ULN, or ≤5.0 x ULN if documented disease involvement of liver
5. Adequate renal function

   a. Creatinine clearance ≥ 50 ml/min (calculated using CKD-EPI formula)
6. Adequate hematologic function a. Platelet count ≥50 x109/L and hemoglobin ≥ 8 g/dL (≥ 80 g/L). Platelet and hemoglobin requirements are independent of transfusions within 7 days of screening assessment and first dose of study drugs.

   b. Absolute neutrophil count ≥ 0.75 x 109/L. Absolute neutrophil count is independent of growth factor support within 7 days of screening assessment and first dose of study drugs.
7. Ability to swallow tablets and comply with outpatient treatment, laboratory monitoring, and required clinic visit for the duration of study participation
8. Women of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (β-hCG) pregnancy test result within 7 days prior to the first dose of study drugs and must agree to use an effective contraception method during the study and for 6 months following the last dose of study drug. Women of non-childbearing potential are those who are postmenopausal greater than 2 year or who have had a bilateral tubal ligation or hysterectomy. Men who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 6 months following the last dose of study drug

Exclusion Criteria:

1. Major surgery within 4 weeks prior to the first dose of study drugs
2. Uncontrolled active systemic infection
3. Known positive serology for human immunodeficiency virus (HIV)
4. Active hepatitis B infection (defined as the presence of detectable HBV DNA, HBe antigen or HBs antigen). Patients with serologic evidence of prior vaccination (HBsAg negative, anti-HBs antibody positive, anti-HBc antibody negative) are eligible. Patients who are HBsAg negative/HBsAb positive but HBcAb positive are eligible, provided HBV DNA is negative and they are willing to take appropriate anti-viral prophylaxis
5. Active hepatitis C infection (defined as detectable hepatitis C RNA in plasma by PCR)
6. Known active cytomegalovirus (CMV) infection. Unknown or negative status are eligible
7. Active, uncontrolled autoimmune phenomenon (autoimmune hemolytic anemia or immune thrombocytopenia) requiring steroid therapy with > 20 mg daily of prednisone or equivalent or for which new therapy was introduced or existing therapy was escalated within the 4 weeks prior to study enrollment to maintain adequate blood counts
8. Clinically significant, uncontrolled cardiovascular disease (≥3 NYHA heart failure, uncontrolled or symptomatic arrythmias), or myocardial infarction within 6 months, or stroke within 6 months, or intracranial bleeding within 6 months prior to start of study drugs
9. Prolongation of the QT interval corrected for heart rate (QTcF) > 470 msec. Note: Patients with QTcF > 470 msec should have EKG repeated. If QTcF again is > 470 msec, then the patient should be referred to cardiology for evaluation. Patient can be enrolled later if cleared by cardiology and repeat QTcF less than 470 msec. QTcF is calculated using Fridericia's Formula (QTcF): QTcF = QT/(RR0.33) a. Correction of suspected drug-induced QTcF prolongation can be attempted at the investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation.

   b. Correction for underlying bundle branch block (BBB) allowed. Note: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker
10. Pregnancy, lactation or plan to breastfeed during the study or within 6 months of the last dose of study treatment
11. Concurrent use of warfarin or another vitamin K antagonist
12. Current treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers. A washout period of at least 5 half-lives of these agents following discontinuation and prior to study entry is required (treatment with moderate CYP3A4 inhibitors or inducers is not excluded)

    a. Because of their effect on CYP3A4, use of any of the following within 7 days of study therapy start or planned use during study participation is prohibited

    i. Grapefruit or grapefruit products

ii. Seville oranges or products from Seville oranges

iii. Star fruit 13. Current treatment with the following P-gp inhibitors: amiodarone, clarithromycin, cyclosporine, erythromycin, ketoconazole, and verapamil. A washout period of at least 5 half-lives of the inhibitor before study entry is required.

14. Known central nervous system involvement by CLL/SLL/RT 15. Active second malignancy unless in remission and with life expectancy > 2 years with exception of patients diagnosed with basal cell or squamous cell carcinoma of the skin or carcinoma "in situ" of the cervix or breast who are eligible even if diagnosed within 2 years. If patients have another malignancy that was treated within the last 2 years, such patients may be enrolled, if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy at MD Anderson Cancer Center, and after consultation with the Principal Investigator.

16. Prior therapy restrictions

a. Cohort 1 (CLL/SLL)

i. Prior receipt of anti-CD20 monoclonal antibody therapy for non-malignant indication, including for autoimmune phenomenon ii. Prior receipt of systemic therapy for CLL/SLL

b. Cohort 2 (RT)

i. Patients who experienced a major bleeding event or grade ≥3 arrythmia on prior treatment with a BTK inhibitor ii. History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor-modified T cell (CAR-T) therapy within 60 days of first dose of study drugs or presence of any of the following, regardless of prior SCT and/or CAR-T therapy timing:

1. Active graft versus host disease (GVHD)
2. Cytopenia from incomplete blood cell count recovery post-transplant
3. Need for anti-cytokine therapy for toxicity from CAR-T therapy or residual symptoms of neurotoxicity > Grade 1 from CAR-T therapy
4. Ongoing immunosuppressive therapy (> 20 mg prednisone or equivalent daily) including GVHD prophylaxis/treatment (calcineurin inhibitors or ruxolitinib)

iii. Patients are required to have the following washout periods prior to planned Cycle 1 Day 1 (C1D1). In addition, prior treatment-related AEs must have recovered to Grade ≤ 1 with the exception of alopecia and Grade 2 peripheral neuropathy.

1. Targeted agents, investigational agents, therapeutic monoclonal antibodies or cytotoxic chemotherapy: 5 half-lives or 2 weeks, whichever is shorter

1. Immunoconjugated antibody treatment within 10 weeks prior to randomization
2. Broad field radiation (≥ 30% of the bone marrow or whole brain radiotherapy) must be completed 14 days prior to study enrollment
3. Palliative limited field radiation must be completed 7 days prior to study enrollment.

   iv. Prior therapy with venetoclax and obinutuzumab is allowed but Richter should not have developed while actively receiving venetoclax or obinutuzumab (active therapy implies having received venetoclax or obinutuzumab within the prior 3 months)

   17. Known hypersensitivity to any component or excipient of study drugs

   18. Malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the study drugs

   19. Receipt of live-virus vaccines within 4 weeks prior to starting study drugs

   20. History of bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2028-04-25 (Estimated); Study Completion 2028-04-25 (Estimated)

PRIMARY OUTCOMES:
The severity of the adverse events (AEs) will be graded according to the U.S. Department of Health and Human Services, National Institutes of Health, National Cancer Institute, Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0. | through study completion an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org